CLINICAL TRIAL: NCT03930108
Title: Validity of Sequential Organ Failure Assessment (SOFA) Score as Predictor of Mortality in Critically-ill Burn Patients
Brief Title: Validity of SOFA Score as Predictor of Mortality in Critically-ill Burn Patients
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, MD, PhD, Anesthesiologist Consultant, Indonesia University
Other Study IDs: IndonesiaUAnes033
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Mortality Prediction
Keywords: Burn injury; Mortality prediction; SOFA score; Organ failure
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mortality outcome
  Interventions: Other: SOFA score

INTERVENTIONS:
Other: SOFA score — Variables of sequential organ failure assessment score, including: P:F ratio; MAP or vasoactive treatment; creatinine or 24-h diuresis; platelet count; serum bilirubin; GCS.

SUMMARY:
SOFA score is valid for mortality predictor for critically-ill patient in high care and intensive care burn unit

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age 18 and above) who admitted to burn unit during sampling period

Exclusion Criteria:

* patients discharged or deceased less than 24 hours of admission
* patients referred to other hospital within 30 days admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical record of adult patients in burn units during a period between January 2012 and December 2017
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2019-02-17 (Actual)

PRIMARY OUTCOMES:
SOFA score Discrimination | 30 days from admission
  SOFA score ability to discriminate outcomes based on variable scores: PaO2/FiO2; MAP/vasoactive treatment; serum creatinine or 24-h diuresis; platelet count; serum bilirubin; GCS
SOFA score Calibration | 30 days from admission
  SOFA score cutoff to predict outcome based on variable scores: PaO2/FiO2; MAP/vasoactive treatment; serum creatinine or 24-h diuresis; platelet count; serum bilirubin; GCS
Correlation between SOFA score variables with outcome | 30 days from admission
  Correlation between patient outcomes with each SOFA score variable: PaO2/FiO2; MAP/vasoactive treatment; serum creatinine or 24-h diuresis; platelet count; serum bilirubin; GCS

SECONDARY OUTCOMES:
Patient outcome | 30 days from admission
  Patient outcome within 30 days of admission to burn units: deceased or survived
SOFA score: Partial Oxygen Pressure (PaO2)/ Fraction of Inspired Oxygen (FiO2) | Day 1
  The score for PaO2/FiO2 variable cutoff:
  0 point for >400 mmHg;
  1. point for <400 mmHg;
  2. points for <300 mmHg;
  3. points for <200 mmHg with respiratory support;
  4. points for <100 mmHg with respiratory support.
SOFA score: Mean Arterial Pressure (MAP) or vasoactive agent usage | Day 1
  The score for MAP or vasoactive agent usage variable cutoff:
  0 point for MAP >=70 mmHg;
  1. point for MAP <70 mmHg;
  2. points for dopamine <= 5 mcg/kg/min OR dobutamine any dose;
  3. points for dopamine >5 mcg/kg/min OR norepinephrine or epinephrine <=0.1 mcg/kg/min;
  4. points for dopamine >15 mcg/kg/min OR norepinephrine or epinephrine >0.1 mcg/kg/min.
SOFA score: Serum creatinine or 24-hour diuresis | Day 1
  The score for serum creatinine or 24-hour diuresis variable cutoff:
  0 point for creatinine <1.2 mg/dL;
  1. point for creatinine 1.2 - 1.9 mg/dL;
  2. points for creatinine 2.0 - 3.4 mg/dL;
  3. points for creatinine 3.5 - 4.9 mg/dL OR diuresis <500 mL/24h;
  4. points for creatinine >5.0 mg/dL OR diuresis <200 mL/24h.
SOFA score: Platelet count | Day 1
  The score for platelet count variable cutoff:
  0 point for >=150 x10^3/mm^3;
  1. point for <150 x10^3/mm^3;
  2. points for <100 x10^3/mm^3;
  3. points for <50 x10^3/mm^3;
  4. points for <20 x10^3/mm^3.
SOFA score: Serum Bilirubin | Day 1
  The score for serum bilirubin variable cutoff:
  0 point for <1.2 mg/dL;
  1. point for 1.2 - 1.9 mg/dL;
  2. points for 2.0 - 5.9 mg/dL;
  3. points for 6.0 - 11.9 mg/dL;
  4. points for >12.0 mg/dL.
SOFA score: Glasgow Coma Scale (GCS) | Day 1
  The score for GCS variable cutoff:
  0 point for 15;
  1. point for 13 - 14;
  2. points for 10 - 12;
  3. points for 6 - 9;
  4. points for <6L.

CONTACTS AND LOCATIONS:
Locations (1):
- Rumah Sakit Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Wardhana A, Basuki A, Prameswara ADH, Rizkita DN, Andarie AA, Canintika AF. The epidemiology of burns in Indonesia's national referral burn center from 2013 to 2015. Burn Open. 2017;1(2):67-73.
- [Background] Queiroz LF, Anami EH, Zampar EF, Tanita MT, Cardoso LT, Grion CM. Epidemiology and outcome analysis of burn patients admitted to an Intensive Care Unit in a University Hospital. Burns. 2016 May;42(3):655-62. doi: 10.1016/j.burns.2015.08.002. Epub 2016 Jan 4. PMID 26762620
- [Background] Taofik S, Senapathi TGA, Wiryana M. Comparison Of Validity Apache II, SOFA And Customized Sequential Organ Failure Assessment (Csofa) For Predicting Non-Surgical Patient. J Anestesiol Indones. 2015;7(2):102-13.
- [Background] Sunaryo A, Redjeki IS, Bisri T. Perbandingan Validasi APACHE II dan SOFA Score untuk Memperkirakan Mortalitas Pasien yang Dirawat di Ruang Perawatan Intensif. Majalah Kedokteran Terapi Intensif. 2012;2(1):11-20.
- [Background] Andrias A, Hanafie A, Wijaya DW. Comparison of APACHE II, SOFA, and CSOFA Scoring System Validity as Mortality Predictor in ICU Patients in H. Adam Malik General Hospital. J Anestesi Perioper. 2017;5(1):17-23j.
- [Background] Bouch DC, Thompson JP. Severity scoring systems in the critically ill. Contin Educ Anaesth Crit Care Pain. 2008;8(5):181-5.
- [Background] Vincent JL, de Mendonca A, Cantraine F, Moreno R, Takala J, Suter PM, Sprung CL, Colardyn F, Blecher S. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998 Nov;26(11):1793-800. doi: 10.1097/00003246-199811000-00016. PMID 9824069
- [Background] Snell JA, Loh NH, Mahambrey T, Shokrollahi K. Clinical review: the critical care management of the burn patient. Crit Care. 2013 Oct 7;17(5):241. doi: 10.1186/cc12706. PMID 24093225
- [Background] Jain A, Palta S, Saroa R, Palta A, Sama S, Gombar S. Sequential organ failure assessment scoring and prediction of patient's outcome in Intensive Care Unit of a tertiary care hospital. J Anaesthesiol Clin Pharmacol. 2016 Jul-Sep;32(3):364-8. doi: 10.4103/0970-9185.168165. PMID 27625487
- [Background] Cardenas-Turanzas M, Ensor J, Wakefield C, Zhang K, Wallace SK, Price KJ, Nates JL. Cross-validation of a Sequential Organ Failure Assessment score-based model to predict mortality in patients with cancer admitted to the intensive care unit. J Crit Care. 2012 Dec;27(6):673-80. doi: 10.1016/j.jcrc.2012.04.018. Epub 2012 Jul 2. PMID 22762932
- [Background] de Brito MR, Barros AG, Valler L, Cardoso FB, Gasparotto AP, Tiziani L, et al. Evaluation of Sequential Organ Failure Assessment (SOFA) Performance in Neurocritical Care Patients Overtime: A Retrospective Cohort Study. J Brain Disord. 2017;1(1):38-43.
- [Background] Nair R, Bhandary NM, D'Souza AD. Initial Sequential Organ Failure Assessment score versus Simplified Acute Physiology score to analyze multiple organ dysfunction in infectious diseases in Intensive Care Unit. Indian J Crit Care Med. 2016 Apr;20(4):210-5. doi: 10.4103/0972-5229.180041. PMID 27303136
- [Background] Cabre L, Mancebo J, Solsona JF, Saura P, Gich I, Blanch L, Carrasco G, Martin MC; Bioethics Working Group of the SEMICYUC. Multicenter study of the multiple organ dysfunction syndrome in intensive care units: the usefulness of Sequential Organ Failure Assessment scores in decision making. Intensive Care Med. 2005 Jul;31(7):927-33. doi: 10.1007/s00134-005-2640-2. Epub 2005 Apr 26. PMID 15856171
- [Background] Lorente JA, Vallejo A, Galeiras R, Tomicic V, Zamora J, Cerda E, de la Cal MA, Esteban A. Organ dysfunction as estimated by the sequential organ failure assessment score is related to outcome in critically ill burn patients. Shock. 2009 Feb;31(2):125-31. doi: 10.1097/SHK.0b013e31817fc3ef. PMID 18650779
- [Background] Karlie J, Wardhana A. External Validation of Belgian Outcome of Burn Injury Score on Burned Patient In Burn Unit Cipto Mangunkusumo General Hospital. New Ropanasuri J Surg. 2017;2(1):90.
- [Background] Emara SS, Alzaylai AA. Renal failure in burn patients: a review. Ann Burns Fire Disasters. 2013 Mar 31;26(1):12-5. PMID 23966893
- [Background] Ibrahim AE, Sarhane KA, Fagan SP, Goverman J. Renal dysfunction in burns: a review. Ann Burns Fire Disasters. 2013 Mar 31;26(1):16-25. PMID 23966894
- [Background] Carson J, Goverman J, Fagan S. Acute renal failure in association with thermal injury. In: Herndon D, editor. Total Burn Care. 5th ed. Elsevier; 2018. p. 318-27.
- [Background] Nielson CB, Duethman NC, Howard JM, Moncure M, Wood JG. Burns: Pathophysiology of Systemic Complications and Current Management. J Burn Care Res. 2017 Jan/Feb;38(1):e469-e481. doi: 10.1097/BCR.0000000000000355. PMID 27183443
- [Background] Enkhbaatar P, Sousse L, Cox R, Herndon D. The pathophysiology of inhalation injury. In: Herndon D, editor. Total Burn Care. 5th ed. Elsevier; 2018. p. 174-83.
- [Background] Marck RE, Montagne HL, Tuinebreijer WE, Breederveld RS. Time course of thrombocytes in burn patients and its predictive value for outcome. Burns. 2013 Jun;39(4):714-22. doi: 10.1016/j.burns.2013.01.015. Epub 2013 Mar 13. PMID 23490002
- [Background] Guo F, Wang X, Huan J, Liang X, Chen B, Tang J, Gao C. Association of platelet counts decline and mortality in severely burnt patients. J Crit Care. 2012 Oct;27(5):529.e1-7. doi: 10.1016/j.jcrc.2011.12.006. Epub 2012 Feb 1. PMID 22300492